CLINICAL TRIAL: NCT00879515
Title: Genetics and Physiology of Social Anxiety in Fragile X
Brief Title: Examining Social, Emotional, and Cognitive Functioning in People With Fragile X and Down Syndromes
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 200210645; K23MH077554 (NIH); DDTR B2-MBA
Record Dates: First submitted 2009-04-09; First posted 2009-04-10 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Anxiety Disorders; Child Developmental Disorders, Pervasive
Keywords: Fragile X Premutation; Fragile X Syndrome; Down Syndrome
MeSH Terms: conditions — Anxiety Disorders; Fragile X Syndrome; Down Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva samples collected at four time periods
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1: Males and females with fragile X syndrome, ages 5 to 25 years old
- 2: Males and females with the FMR1 premutation, ages 5 to 25 year old
- 3: Males and females with Down syndrome, ages 5 to 25 years old
- 4: Males and females with normal development, ages 5 to 25 years old

SUMMARY:
By testing physiological responses to anxiety in people with nervous system developmental disorders, this study will identify specific physiological characteristics associated with response to anxiety treatments.

DETAILED DESCRIPTION:
Anxiety is a common and significant problem for people suffering from disorders of nervous system development, including fragile X syndrome. There are few validated treatments for anxiety in people with these disorders, in part because the biological basis of anxiety in neurodevelopmental disorders has not been clearly described. This study will evaluate the physiological responses of people with fragile X syndrome, Down syndrome, and the fragile X premutation (a mild version of the genes that cause fragile X syndrome) to a variety of sensory, emotional, and social stimuli. By analyzing the data collected for this study, researchers aim to identify physiological characteristics linked to subgroups within the disorders, demonstrate links between physiological responses and behavioral or psychiatric symptoms, and measure physiological changes in people receiving treatment for their disorders.

Participation in this study will include one testing session, which will take between 3 and 3.5 hours. Participants who receive treatment for their anxiety may be asked to complete this testing a second time, after their treatment. During the testing session, sensors will be placed on participants' skin in several locations to measure heart rate, sweat response, and eye-blinks. Participants will then be asked to respond to multiple stimuli: sounds, lights, smells, pictures that elicit different types of emotions, an interaction with an unfamiliar person, and specialized toys. In addition, participants will undergo blood testing and have several samples of their saliva collected on the day of the testing session. Participants will also be asked to collect additional saliva samples at home three times a day on 4 different days. Child participants and their parents may also be asked to complete questionnaires and interviews about behavioral and emotional problems.

ELIGIBILITY:
Inclusion Criteria:

* Fragile X premutation or fragile X syndrome, measured by DNA testing; Down syndrome, confirmed by chromosomal analysis; or normally developing control
* Normal hearing

Ages: 5 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Individuals with fragile X syndrome, Down syndrome, the fragile X premutation, and normal development
Sampling Method: Non-Probability Sample
Enrollment: 511 (Actual)
Dates: Start 2005-10; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Fear-potentiated startle reflex | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- M.I.N.D. Institute, University of California, Davis, Sacramento, California, United States

REFERENCES:
- See also: Click here for more information about the M.I.N.D. Institute — http://www.ucdmc.ucdavis.edu/mindinstitute/